CLINICAL TRIAL: NCT01975051
Title: A Study to Explore Association of Treatment Regimens for Visceral Leishmaniasis, Host Immunological, Genetical and Nutrition Factors With Post-kala-azar Dermal Leishmaniasis (PKDL)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: University of Nagasaki. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PR-12057
Record Dates: First submitted 2013-10-23; First posted 2013-11-04 (Estimated); Last update posted 2014-11-05 (Estimated); Status verified 2012-11

CONDITIONS: Post-kala-azar Dermal Leishmaniasis
Keywords: Kala- azar; PKDL; Treatment; Pathogenesis; Bangladesh
MeSH Terms: conditions — Leishmaniasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Miltefosine (Experimental): Tablet Miltefosine 100 mg daily in two divided doses for 12 weeks.
  Interventions: Drug: Mitefosine

INTERVENTIONS:
Drug: Mitefosine — Tablet Miltefosine 100 mg in two devided doses for 12 weeks
  Other Names: Brand name: Impavido

SUMMARY:
We hypothesize that PKDL develop after SSG as well as after Miltefosine mono-therapy for VL; anti-inflammatory cytokines such as IL-10, TGF-β, serum lipids play key role for its pathogenesis & PKDL patients are genetically predisposed; diagnostic tool based on immunofluorescence technique will be more sensitive than slit skin examination for diagnosis of PKDL.

DETAILED DESCRIPTION:
Background:Post-kala-azar dermal leishmaniasis is a skin disorder caused by the Leishmania donovani and usually develops after treatment for visceral leishmaniasis. The public health importance of this condition is that it plays as an inter-epidemic reservoir of visceral leishmaniasis.It is believed that the condition is associated with sodium stibogluconate (SSG) monotherapy for visceral leishmaniasis; however evidence is lacking to support this. Further no study has been carried out to explore the pathogenesis of PKDL in Bangladesh. Also no information is available related to development of PKDL after treatment of VL with miltefosine monotherapy in Bangladesh.Better knowledge on pathogenesis of PKDL will help to predict and design intervention to prevent the development of PKDL. This will help to reduce the numbers of inter-epidemic reservoir for VL and hence will contribute to the national kala-azar elimination program.

Objectives:1. To investigate the incidence of PKDL after SSG or Miltefosine mono-therapy for VL; 2. To investigate serum level of IL-10, TGF-β and markers of lipid metabolism (serum cholesterols) before and after treatment of PKDL; 3. To investigate the mRNA expression of IL-10, TGF-β in skin lesion of PKDL; 4. To investigate the association of gene polymorphism of IL-10, TGF-β and PKDL; 5. To develop a new diagnostic tool for diagnosis of PKDL by detection of LD antigen in the skin tissue by punch biopsy using immunofluorescence technique; and, 6. To investigate leishmania antigens and anti-leishmania antibodies in urine before and after treatment of PKDL and evaluate possibility to use them as diagnostic tools.

Methods:1. The incidence of PKDL after treatment for VL will be investigated through studying a retrospective cohort which will be identified by cross-sectional survey; 2. serum level of cytokines and lipid profile will be measured respectively by cytometric bed-array and autoanalyzer before and after treatment for PKDL; 3. mRNA expression of cytokines will be measured real-time PCR before and after treatment for PKDL; 4. gene polymorphism will be investigated by DNA sequencing; 5. the new diagnostic tool will be developed using immunofluorescence technique; and, 6. urine antigens and antibodies will be detected by ELISA.

ELIGIBILITY:
Inclusion Criteria:

* History of Visceral Leishmaniasis
* Presence of hypopigmented rash
* Rk39 strip test positive
* Written informed consent from the participant

Exclusion Criteria:

* Any medical condition that may affect the safety of the patient during study procedure
* Any condition which comprises the ability to comply the study procedure
* Presence of splenomegaly
* Posotive skin smear for mycobacterium leprae
* Positive skin smear for fungus
* Pregnancy test positive

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2013-01; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Explore the association of treatment regimens for visceral leishmaniasis, host immunological, genetical and nutrition factors with Post-kala-azar Dermal Leishmaniasis (PKDL) | Three years
  1. PKDL burden among VL patients treated with SSG and miltefosine in the past; 2. Association of serum level of IL-10, TGF-β and serum level of cholesterols before and after treatment of PKDL; 3. mRNA expression of IL-10, TGF-β in skin lesion before and after treatment; 4. association of gene polymorphism of IL-10, TGF-β and PKDL; 5. diagnostic sensitivity of immunofluorescence technique compared to skin slit examination and PCR; and, 6. titer of urine antigens and antibodies before and after treatment of PKDL.

CONTACTS AND LOCATIONS:
Overall Officials: Dinesh Mondal, MB; MD; PhD, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- Dinesh Mondal, Dhaka, Dhaka Division, Bangladesh